CLINICAL TRIAL: NCT03052374
Title: Video-Feedback Interaction Guidance for Improving Interactions Between Depressed Mothers and Their Infants ("VID-KIDS")
Acronym: VID-KIDS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Nicole Letourneau, Professor of Nursing, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB-Ethics ID #: REB16-1811
Record Dates: First submitted 2017-02-02; First posted 2017-02-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Post Partum Depression
Keywords: Video-Feedback Interaction Guidance; Depressed Mothers and their Infants
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Mothers will receive standard care such as referral to psychotherapy (intervention mothers will have the same access) over the same length of time.
- VID-KIDS Intervention Program Group (Experimental): RN review photos of infant engagement/disengagement cues. NCAST Teaching Activity, mothers asked to perform task advanced for infant's level, recorded. 1st-View, no feedback, mothers reveal infant cues. RN records infant/mother's response, later discussion. 2nd, RN and mother co-view interaction with time for replay/review parts of sensitivity and responsiveness. RN feedback: praising desired maternal behaviours; information on infant cues; maternal response to infant distress; and use of cognitive growth fostering language. 3rd, all concepts discussed in past views, use positive reinforcement to affirm aspects of sensitivity, useful feedback for areas of growth. Post-Debrief, RN and mother discuss interests of the mother. Mothers encouraged to note infants' engagement/disengagement cues.
  Interventions: Behavioral: VID-KIDS Intervention Program

INTERVENTIONS:
Behavioral: VID-KIDS Intervention Program — Investigators created VID-KIDS for mothers with PPD to improve sensitivity and positive responsiveness towards their infants. Video-feedback has the advantage of being visually concrete yet "distant" because the action and the feedback are not concurrent; this helps mothers maintain an element of objectivity that may minimize guilty feelings associated with potential perceived lack of parenting skills. Video-feedback interventionists are trained by investigators with manualized modules. Including: Introduction to Video-feedback; NCAST Keys to Caregiving Program; Infant Engagement and Disengagement Cues; Video-feedback Intervention Protocol; Overview of Behaviours of Interest; Case Studies; and Examples of Strengths-Based Feedback. VID-KIDS intervention follows an 8-step protocol.
  Other Names: NCAST Program
  Arms: VID-KIDS Intervention Program Group

SUMMARY:
Postpartum depression (PPD) is a major public health issue. Known as "the thief that steals motherhood" since symptoms obstruct a mother's capacity for understanding and enjoying her baby, PPD affects approximately 1 in 5 moms. Built via "serve and return" interactions (e.g. baby smiles, mom smiles back), sensitive and responsive exchanges are the foundation for healthy child development but are diminished by PPD, resulting in interactions that place children at risk for behavioural and cognitive problems. Infants perceive PPD as stressful; stressors stimulate the brain's hypothalamic pituitary adrenal axis (HPA) and trigger stress hormone (cortisol) release, which, in turn, negatively affects developing infant brains by decreasing brain volume. Infants' critical periods of brain development are vulnerable to long-term effects of cortisol, explaining some of the problematic developmental outcomes observed in children of depressed mothers.

How can the investigators support depressed mothers and their infants? Successfully treating PPD does not always benefit mother-child relationships; however, this research builds on a successful pilot that demonstrated that nurse-guided video feedback improved mother-infant interactions in the context of PPD. By improving interaction quality, depressed mothers may be motivated to engage in more play and, in turn, infants who appear interested and ready to interact are more likely to elicit positive, enjoyable experiences from mothers. Building on the pilot, the investigators will trial the effectiveness of VID-KIDS (Video-Feedback Interaction Guidance for Improving Interactions Between Depressed Mothers and their Infants) on maternal-infant interaction and infant cortisol patterns as well as infant development, maternal symptoms of depression and anxiety, and parenting self-efficacy. If successful, future aims are to 1) integrate VID-KIDS into existing services of Calgary Public Health; and 2) commercialize VID-KIDS for dissemination.

DETAILED DESCRIPTION:
Background & Rationale: Affecting ~19% of mothers, postpartum depression (PPD) reduces maternal sensitivity and positive responsiveness to infant cues and bids for caring attention. Infants perceive these behaviours as stressful which stimulates the hypothalamic pituitary adrenal axis, triggering cortisol release which, at persistently elevated levels, inhibits neurogenesis during critical periods of brain development. Elevated infant cortisol of infants of mothers with PPD may explain later poor child cognitive development and hyperactivity and anxiety problems into adolescence. The negative developmental outcomes from poor quality interactions and disrupted cortisol patterns underscores the urgency for intervening. Treating PPD successfully, has not consistently improved maternal-infant (M-I) interaction quality and children's development. Parent training promoting sensitive, responsive interactions may help infants of depressed mothers develop optimally.

Research Question & Objectives: Conduct a randomized controlled trial (RCT) with depressed mothers of infants aged 2-6 months designed to alter negative M-I interaction and child development associated with PPD. Objective: examine effect of the intervention, VID-KIDS ("video-feedback intervention to promote improved interactions between mothers and their kids"), on: 1) M-I interaction; 2) infant cortisol patterns, infant development, maternal symptoms of PPD, anxiety, and parenting stress. Anticipate to improve: 1) M-I interactions and infant development, infant cortisol; 2) symptoms of PPD, anxiety, parenting stress, and infant development. The investigators will conduct cost-benefit analyses.

An additional objective is to collect infant buccal cells for future genetic/epigenetic analyses. Research has suggested biological sensitivity, assessed via genotyping specific genetic variants and alleles may confound effects of interventions of this nature. Intervention may affect the epigenome, particularly the number or nature of methylated DNA sites, of treated infants differently than untreated infants that may link to infant development. This portion of the study is optional for parents-they can opt out of buccal cell collection.

Methods: The study will implement a parallel group RCT compared to resource and referral program (standard care) for mothers with PPD and their infants. After baseline assessment, over the following 9-weeks, mothers randomized to the intervention will receive 3-video-feedback sessions during home visits conducted at 3-week intervals. Mothers randomized to the control condition will receive standard care. Both groups will be assessed at baseline, immediately following the 9-week treatment/standard care interval (post-test), then 2-months later (delayed post-test).

Both control and intervention mothers will have access to standard care over the study period. Mothers' use of such health services will be documented. The investigators will adhere to CONSORT guidelines.

Intervention description. Video-feedback interventionists will be trained by Co-PI Tryphonopoulos using a manualized curriculum of 7-themed modules offered in a 4-day workshop. Training modules will include: 1) Introduction to Video-feedback; 2) NCAST Keys to Caregiving Program; 3) Infant Engagement and Disengagement Cues (using NCAST's BabyCues: A Child's First Language Cards®; 4) Video-feedback Intervention Protocol; 5) Overview of Behaviours of Interest; 6) Case Studies; and 7) Examples of Strengths-Based Feedback.

The intervention follows an 8-step protocol:

Ice-breaking. Interventionist initiates rapport with the participant.

Overview of Infant Engagement and Disengagement Cues. Using NCAST's BabyCues, interventionists review coloured photo cards that illustrate and explain the behavioural cues commonly seen in infants, including potent and subtle engaging and disengaging cues.

NCAST Teaching Activity. Using the Nursing Child Assessment Teaching Scale (NCATS) protocols and elements, mothers are asked to perform a teaching task more advanced than their infant's age level.

Recording Interaction. Mothers and infants are observed and video-recorded.

Initial-Viewing. Specific feedback is not provided during the initial viewing. Mothers are asked to reflect on and point out any infant cues they recognize. Interventionist documents the presence or absence of infant cues and mother's response for later discussion.

Second-Viewing. Interventionist and mother co-view the recorded interaction with opportunities provided for replay/slow review portions emphasizing sensitivity and responsiveness. Interventionist provides feedback: using praise reinforcing desired maternal behaviours; information on infant cues; appraisal of maternal response to infant distress; and use of cognitive growth fostering language.

Third-Viewing. The final viewing, integrates all of the concepts discussed in the previous screenings, using positive reinforcement to emphasize optimal aspects of sensitivity, responsiveness and constructive feedback suggesting areas for growth.

Post-viewing Debrief. Interventionist and mother conclude the video-feedback session discussing whatever interests the mother. Mothers are encouraged to make note their infants' engagement/disengagement cues and responses to these non-verbal behaviours.

Video feedback sessions last 60-90min. Subsequent sessions follow same protocol (new teaching activities) and build on the previous interaction guidance discussions.

ELIGIBILITY:
Inclusion Criteria:

* Recruitment will be conducted through Calgary Public Health's immunization program. Public Health RNs routinely screen mothers for PPD during infants' vaccination clinic appointments using the Edinburgh Postnatal Depression Scale (EPDS) at 2, 4, and 6 months of age. EPDS scores>12 are indicative of probable major depression with postpartum onset and make a mother eligible for our study. Approximately 500 mothers per year (40/month) screen >12 on the EPDS. The investigators have agreed to support a part-time Calgary Public Health staff person to review screening records and contact potential participants to determine if they are willing to be contacted by a the VID-KIDS Project Manager for further information about the study. If mothers agree, then the VID-KIDS Project Manager will contact the mother to explain the study, further assess eligibility, and if appropriate conduct the informed consent procedure.

If the investigators are able to successfully invite 40% of these mothers, then the investigators project that the investigators will be able to recruit at least 16 participants per month, giving us our sample in 20-24 months. Since the inception rate of PPD is greatest within the first 12 weeks of delivery, screening mothers at these strategic intervals is particularly advantageous. Moreover, Co-I McNeil and Collaborator Philley (Director of Research and Director of Nursing, Calgary Public Health, respectively) have successful experience with this feasible approach. Eligibility will be based on 1) a cut-off of greater than 12 (indicating probable PPD) on the Edinburgh Postnatal Depression Scale (EPDS) 20; and 2) infant aged 2-6 months at baseline. Mothers will not be excluded for taking anti-depressants or using other interventions for PPD (i.e., counseling, psychotherapy). However, mothers who are receiving other parenting services (e.g., Circle of Security program, infant-parent psychotherapy) will be excluded.

Exclusion Criteria:

* None as long as they meet Inclusion Criteria

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be new mothers suffering from PPD
Enrollment: 400 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
NCAST assessment scale will be used to evaluate Mother-Infant (M-I) interactions | through study completion, an average of 18 weeks
  Using the Nursing Child Assessment Satellite Training (NCAST) assessment scale will be used to evaluate Mother-Infant (M-I) interactions. See Study Detailed Description and intervention arm for more information on the NCAST Program.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Letourneau, RN, PhD, Principal Investigator — University of Calgary
Locations (1):
- Maternal Newborn Child and Youth Strategic Clinical Network, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Informed Consent Form — http://childstudies.ca/contact
- Available data/document: Study Protocol — http://childstudies.ca/contact
- Available data/document: Statistical Analysis Plan — http://childstudies.ca/contact